CLINICAL TRIAL: NCT06537830
Title: Validity And Reliability of Wearable Motion Sensors in Knee Joint Range of Motion Measurement
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Other Study IDs: Acetinkaya004
Record Dates: First submitted 2024-07-28; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Range of Motion; Knee
Keywords: Wearable motion sensors; MetamotionRL; IMUs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: The aim of this study is to examine the validity and reliability of a wearable motion sensor, which is an inertial measurement units (IMUs) sensor, in measuring knee joint active flexion movement angles.

Methods: The study included 70 Health Sciences Faculty students between the ages of 18-25. The dominant knee joint range of motion of the participants was measured by two raters with a digital goniometer (Meloq EasyAngle) and wearable motion sensors (MetaMotionRL). A 10-minute rest was given between each measurement. The data were analyzed using the IBM® SPSS® Statistics for Windows software (Version 27.0). Mean ± standard deviation (Mean ± SD) and percentage (%) were used for the descriptive variables. Intra- and inter-rater reliability was tested with intraclass correlation coefficient (ICC) and Bland-Altman analysis. ICC values less than 0.5 were classified as poor, values between 0.5 and 0.75 as moderate, values between 0.75 and 0.9 as good, and values greater than 0.90 as excellent reliability. Paired samples t test was used to compare test-retest measurements. Concurrent validity was determined by Pearson correlation coefficient. The significance value was accepted as p<0.05.

DETAILED DESCRIPTION:
Before knee range of motion measurements, all participants were given verbal information about the measurements. Participants were asked to wear shorts that exposed their knees. While the participants were lying in the prone position on the examination table, their dominant knee range of motion was measured with both EasyAngle and MetaMotionRL by two different physiotherapists.

EasyAngle digital goniometer and universal goniometer measurement results were compared and it was concluded that EasyAngle is a valid and reliable evaluation tool.

MetaMotionRL (MBientlab Inc., San Francisco, USA); Includes 9-axis inertial measurement units and environmental monitoring sensor. It features gyroscope, accelerometer, magnetometer and sensor fusion. Real-time communication is provided via BluetoothLE. Data can also be saved to 8 megabyte NOR flash memory. There are free, open-source applications and applications for fast data collection.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-25
* volunteering to participate in the study

Exclusion Criteria:

* a history of orthopedic surgery or trauma to the lower extremity
* knee pain felt during joint range of motion measurement
* inability to maintain a prone position

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Seventy healthy student were included between December 2021 and April 2022, the study was approved by Haliç University Non-Invasive Ethics Committee (173/01.12.2021). All participants completed written informed consent. Seventy healthy students (40 female, 30 male) from Haliç University Faculty of Health Sciences were included in the study.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Digital goniometer measurement | at baseline
  Participants were asked to wear shorts that exposed their knees. While the participants were lying in the prone position on the examination table, their dominant knee range of motion was measured with EasyAngle (Meloq©, Stockholm, Sweden) digital goniometer by physiotherapists (rater I). The participant was instructed to bend his knee and bring his heel as close to his hip as possible. The degree of dominant knee active flexion was measured three times by the rater I with a EasyAngle (Meloq©, Stockholm, Sweden) digital goniometer (the pivot point was determined as the lateral epicondyle of the femur), and the highest value was recorded.
MetaMotionRLs measurement | at baseline
  Two MetaMotionRLs were fixed to the lateral thigh and leg with velcro strap, at the level of the midpoint of the tibia and femur in the dominant lower extremity by the rater I. Two MetaMotionRL motion sensors were used simultaneously. MetaMotionRL was used by connecting via Bluetooth with the free MetaROM (application) smart phone application. The participant was asked to flex his knee as much as possible. Three measurements were made and the highest value shown in the app was recorded. Following this, the sensors were removed and placed again after 10 minutes and measured a second time by the same rater using the same method, the highest value was recorded. Following removal of the sensors, the participant was taken to a different examination table in the same room. And the rater II placed the sensors and repeated the MetaMotionRL measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Güneş Yavuzer, Prof., Study Director — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No